CLINICAL TRIAL: NCT06202781
Title: Using Single-cell Sequencing to Explore Tumor Microenvironment in Gastric Cancer Patients Treated With Combined Immunotherapy and Chemotherapy
Brief Title: Tumor Microenvironment in Gastric Cancer Patients Treated With Combined Immunotherapy and Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xinxin Wang, Prof., Chinese PLA General Hospital
Other Study IDs: scgc1
Record Dates: First submitted 2024-01-01; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer; Tumor Microenvironment; Immunotherapy; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pre-treatment: Advanced gastric cancer patients prior to receiving combined immunotherapy and chemotherapy
  Interventions: Drug: SOX plus PD-1 inhibitor; Procedure: Gastroscopic biopsy
- Post-treatment: Advanced gastric cancer patients who have received 2 to 8 cycles of combined immunotherapy and chemotherapy
  Interventions: Drug: SOX plus PD-1 inhibitor; Procedure: Gastroscopic biopsy
- Response: Advanced gastric cancer patients who have achieved complete response (CR) or partial response (PR) after receiving combined immunotherapy and chemotherapy
  Interventions: Drug: SOX plus PD-1 inhibitor; Procedure: Gastroscopic biopsy
- Non-response: Advanced gastric cancer patients who have achieved stable disease (SD) or progressive disease (PD) after receiving combined immunotherapy and chemotherapy
  Interventions: Drug: SOX plus PD-1 inhibitor; Procedure: Gastroscopic biopsy

INTERVENTIONS:
Drug: SOX plus PD-1 inhibitor — S-1, Oxaliplatin and nivolumab/sintilimab
Procedure: Gastroscopic biopsy — Gastroscopy and biopsy

SUMMARY:
The goal of this study is to analyze the tumor microenvironment (TME) in gastric cancer patients treated with combined immunotherapy and chemotherapy. The main questions it aims to answer are:

* Provide profiles of TME between pre-treatment and post-treatment to gain insights into the mechanisms of immunotherapy combined with chemotherapy in advanced gastric cancer
* Investigate the crucial factors affecting treatment efficacy by comparing gastric cancer patients with varying treatment responses

ELIGIBILITY:
Inclusion Criteria:

* Non-bedridden, aged 18 to 70 years old;
* Eastern Cooperative Oncology Group (ECOG) score is 0 to 1;
* Histologically confirmed gastric adenocarcinoma with evaluable lesions based on RECIST 1.1;
* Advanced gastric cancer;
* Ready for receiving S-1 plus oxaliplatin chemotherapy and either nivolumab or sintilimab

Exclusion Criteria:

* History of other malignant diseases in the last 5 years;
* Prior chemotherapy, radiotherapy or immunotherapy;
* Not receiving S-1 plus oxaliplatin chemotherapy and either nivolumab or sintilimab.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced gastric cancer patients receiving S-1 plus oxaliplatin chemotherapy and either nivolumab or sintilimab
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Single-cell profiling | 6 months
  Single-cell transcriptome and immune repertoire sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China